NCT number: NCT02488291

**Document date:** June 2016

Funds: None

Table 1. Characteristics of parturients in labour analgesia

| Monitored Variables | Ropivacaine Sufentan<br>(n=30) (n=30) | | t | P |
|---|---|---|---|---|
| Age (yr) | 29.17±2.49 29.40±3.54 | | -0.295 | 0.769 |
| Height (cm) | 162.1±5.07 | 162.1±5.07 161.9±5.12 | | 0.900 |
| Weight (kg) | 67.0±7.19 | 67.9±7.62 | -0.523 | 0.603 |
| active stage (min) | (min) 393.7±139.07 363.93±157. | | 0.775 | 0.441 |
| Second stage of labor (min) | 64.30±39.21 | 69.67±34.68 | -0.561 | 0.577 |
| Gestational Weeks (week) $38.83 \pm 0.9$ | | 38.93 ±1.05 | -0.394 | 0.695 |

Data represent mean  $\pm$  SD, there were no significant changes in age, height, weight, gestational weeks, actice stage and second stage of labor between two groups. Statistical analysis was performed by using paired t-test.

Table 2 Side effect and VAS score for two groups (n=30)

| Complications and VAS | Ropivacaine (n=30) | Sufetanil<br>(n=30) | x <sup>2</sup> /t | P |
|---|---|---|---|---|
| Nausea and vomiting/n(%) | 5 (16.7) | 4(13.3) | 0.131 | 0.718 |

| Pruritus/n(%) | 1 (3.3) | 1(3.3) | - | - |
|---|---|---|---|---|
| Hypotension/n(%) | 0 0 | | - | - |
| Respiratory depression/n(%) | 0 | 0 | - | - |
| VAS Before labor analgesia | 8.13±1.76 | 8.33±1.27 | -0.360 | 0.721 |
| VAS for 30 min after labor analgesia | 2.70±1.77#### | 2.80±1.56#### | -0.232 | 0.817 |
| VAS for 60 min after labor analgesia | 1.37±1.54#### | 1.53±1.61#### | 0.140 | 0.889 |
| VAS for Full dilatation of cervix | 3.53±2.05#### | 3.83±1.68#### | -0.809 | 0.422 |
| VAS for Fetal delivery | 2.80±1.88#### | 3.30±1.62#### | -0.759 | 0.452 |

All data are shown as number or mean  $\pm$  SD, \*\*\*\* Significantly different compared with VAS before labor analgesia (P < 0.0001). Statistical analysis was performed by using paired t-test in comparison to Sufetanil group.

Table 3 Maternal and fetal hemodynamic data for two groups (n=30)

| Group | Different<br>time<br>points | Systolic<br>pressure /<br>mmHg | Diastolic<br>pressure /<br>mmHg | Heart rate /<br>bpm | Fetal heart rate / bpm |
|---|---|---|---|---|---|
| Ropivacaine | Before labor analgesia | 124.50±13.43 | 76.17±7.81 | 84.00±12.80 | 141.07±9.43 |
| | 60 min after<br>labor<br>analgesia | 119.37±9.01 | 72.50±6.65 | 79.83±13.06 | 138.87±8.94 |
| Sulfetanil | Before labor analgesia | 120.57±13.41 | 73.93±9.55 | 81.00±11.17 | 136.83±10.61 |
| | 60 min after<br>labor<br>analgesia | 116.89±12.80 | 71.21±9.32 | 78.00±11.35 | 135.79±10.10 |

Statistical analysis was performed by using paired t-test in comparison to

Sufetanil group. There were no significant change between two groups (P > 0.05).